CLINICAL TRIAL: NCT04917978
Title: Association of Hb F Level With Clinical Severity of Beta Thalassemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: ZhuHai Hospital (Other); Shenzhen Children's Hospital (Other Government); Shenzhen Second People's Hospital (Other); Jiangmen Maternity and Child Health Care Hospital (Unknown); Yongzhou Maternity and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: HbF-Beta thalassemia
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Beta Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- beta thalassemia patients
  Interventions: Diagnostic Test: Hematological Phenotype Analysis

INTERVENTIONS:
Diagnostic Test: Hematological Phenotype Analysis — Hematological parameters were determined with an automated hematology analyzer (Sysmex, Japan), and hemoglobin analysis was performed with either high-performance liquid chromatography (Bio- Rad, USA) or capillary electrophoresis (Sebia, France and Helena, USA).

SUMMARY:
The production of Hb F after birth is an important factor in modifying the clinical severity of beta thalassemia because an increased gamma-globin level will bind the additional a-globin and form Hb F. The objective of this project is to evaluate the association of Hb F level with phenotypic diversity of patients with beta thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with beta-thalassemia

Exclusion Criteria:

* Iron Deficiency Anemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: β-thalassemia patients from Southern China
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Hb F level and severity of anemia | 3 years
  Observational study that analyzed association of Hb F level and anemia severity in patients

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China